CLINICAL TRIAL: NCT03679078
Title: An Evaluation of the Tolerance, Compliance, Acceptability and Safety of a New Oral Nutritional Supplement in Dysphagic Patients
Brief Title: IDDSI Nutritional Drink for Dysphagia Study
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Project suspended whilst intervention is updated
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IDDSIL2
Record Dates: First submitted 2018-08-29; First posted 2018-09-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dysphagia; Malnutrition
MeSH Terms: conditions — Deglutition Disorders; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IDDSI nutritional supplement drink (Experimental): Single arm designed, 28day on IDDSI nutritional supplement drink
  Interventions: Dietary Supplement: IDDSI nutritional supplement drink

INTERVENTIONS:
Dietary Supplement: IDDSI nutritional supplement drink — ready-to-use nutritional supplement drink to be taken daily for 28 days

SUMMARY:
This study will evaluate the gastrointestinal (GI) tolerance, compliance , acceptability and safety of a ready-to-use oral nutritional supplement drink for patients with dysphagia.

DETAILED DESCRIPTION:
Dysphagia is a complex condition common in a number of diagnoses including stroke, Parkinson's disease, head and neck cancer, dementia, learning disabilities and gastric/oesophageal motility disorders.

A modified textured diet and/or fluid is considered as an effective intervention in management of dysphagia. The International Dysphagia Diet Standardisation Initiative (IDDSI) have developed a new framework around the terms and descriptors used in the management of individuals with dysphagia. Malnutrition is very common in patients with dysphagia and the use of pre-thickened oral nutritional supplements (ONS) has been found as an effective way to manage this. However, due to impairment in the swallow process, dysphagic patients require pre-thickened oral nutritional supplement to ensure safe consumption of these nutritional supplements.

40 participants, requiring a new pre-thickened oral nutritional supplement in line with the new IDDSI framework recruited from hospitals, outpatients clinics, care homes, community hospitals, community dietetic/speech and language therapy services or stroke rehabilitation units will receive the ready-to-use oral nutritional supplement for a 4 week intervention period. This study aims to primarily evaluate gastro-intestinal tolerance, with secondary outcomes including compliance, acceptability, nutrient intake, anthropometry and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years
* Patients with a requirement for ≥ 250kcal/day from a milkshake style ONS for ≥ 4 weeks or current users of ONS
* Patients identified to require mildly thick (IDDSI level 2) fluids.
* Patients competent to provide written informed consent and able to answer questions
* Patients able to take study ONS orally

Exclusion Criteria:

* Patients that lack capacity to provide informed consent
* Patients that are unable to take study ONS orally
* Participants with chronic renal disease requiring dialysis
* Participants with liver failure
* Participants that are pregnant or lactating
* Participation in other studies that may interfere with this study
* Participants receiving 100% total nutritional requirements from tube feeding or parenteral nutrition
* Patients with galactosaemia or lactose intolerance
* Patients receiving palliative or end of life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance | Day 1, Day 2, Day 3, Day 10, Day 17, Day 24 and Day 31
  Gastro-intestinal tolerance will be assessed daily throughout a 3 day baseline period before starting the study ONS and at the end of each week (day 10, day 17, day 24, day 31) using a standardised GI tolerance questionnaire including questions on number of bowel movements per day, other gastrointestinal symptoms such as flatulence, bloating, burping and abdominal discomfort. Patient-reported gastrointestinal symptoms with scale range for each symptom as s scale range minimum = none, maximum = severe.
  Change of symptom from baseline scale minimum = no change, maximum = worse.

SECONDARY OUTCOMES:
Compliance | Once during baseline period (Day 1) and then daily through intervention period (Days 4-31)
  Daily questionnaire on amount of nutritional drink prescribed and amounts actually consumed. Amount of daily ONS actually consumed scale minimum = 0%, maximum = 100%
Acceptability: Brief tick-box questionnaire | Day 1, Day 17, Day 31
  Brief tick-box questionnaire on overall liking and acceptability of product, including texture and feel of nutritional drink, flavor and ease of use. Scale minimum = dislike very much, maximum = like very much Scale minimum = very inconvenient, maximum = very convenient Scale minimum = very difficult, maximum = very easy
Anthropometry | Day 1 and Day 31
  Measurements of height and weight with Body Mass Index (BMI) calculated at baseline and end of study.
Nutrient intake | Day 1, Day 17 and Day 31
  Three dietary recalls relating to the the past 24 hours of Day 1, Day 17 and Day 31 to capture all food and fluids consumed. This will subsequently be analysed in dietary software.
Safety (Adverse events reporting) | 31 days.
  Reporting of any adverse events that occur throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, Dr, Study Director — Nutricia Ltd UK
Locations (8):
- United Kingdom (8):
  - Aneurin Bevan University Health Board, Caerleon
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Dudley Group NHS Trust, Dudley
  - Cwm Taf University Health Board, Llwynypia
  - Croydon Health NHS Trust, London
  - Lewisham and Greenwich NHS Foundation Trust, London
  - Great Western Hospitals NHS Foundation Trust, Swindon
  - Weston Area Health Trust, Weston-super-Mare

IPD SHARING:
Plan to Share IPD: No